CLINICAL TRIAL: NCT04364971
Title: Comparison of Multiradius and Singleradius Prosthesis Design in Total Knee Arthroplasty Using With Association Sagittal Patellar Offset and Anterior Knee Pain
Brief Title: Comparison of Multiradius and Singleradius Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Orkhan Aliyev, Resident Doctor, Department of Orthopaedics and Traumatology, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 259486
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Gonarthrosis; Primary; Gonarthrosis; Gonarthrosis; Primary, Bilateral; Knee Osteoarthritis; Knee Arthritis
Keywords: multiradius; singleradius; total knee arthroplasty; sagittal patellar offset; anterior knee pain
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- singleradius (Experimental): Single Radius(SR) femoral design will be perfomed to patients who is going to total knee arthroplasty. Single Radius femoral design is one of knee prosthesis' pattern which shows variation in knee kinematics
  Interventions: Procedure: singleradius and multiradius total knee arthroplasty
- Multiradius (Experimental): Multi Radius(MR) femoral design will be perfomed to patients who is going to total knee arthroplasty. Multi Radius femoral design is one of knee prosthesis' pattern which shows variation in knee kinematics
  Interventions: Procedure: singleradius and multiradius total knee arthroplasty

INTERVENTIONS:
Procedure: singleradius and multiradius total knee arthroplasty — singleradius and multiradius total knee arthroplasty

SUMMARY:
The Investigators would like to compare multiradius and single-radius total knee arthroplasty using with association between sagittal patellar offset and anterior knee pain in subjects having undergone bilateral total knee replacement.

DETAILED DESCRIPTION:
A prospective, interventional study. A total of to 494 subjects requiring bilateral multiradius( n=247) and singlerasius(n=247) knee arthroplasty will be enrolled. Anterior femoral offset, femoral diameter and patellar offset will be measured by orthopaedic surgeons. In addition, Visual Analogue Scale Score, Oxford Knee Score, WOMAC, SF12 and SF36 will be evaluated postoperative in patients long-term follow up to see if there is a relationship between anterior femoral offset and anterior knee pain. In the direct lateral knee joint radiograph, the distance between the two parallel axis extending from both cortices of the femur is measured as "femoral diameter".The remaining length between the anterior axis and the maximum peak at the anterior of the prosthesis is considered as an "anterior femoral offset". Sagittal patellar offset is accepted by us as the ratio of the anterior femoral offset to the remaining distance between the maximum anterior point of the patella and the posterior vertex in the direct lateral knee joint radiography.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of end-stage primary gonarthrosis

Exclusion Criteria:

* History of malignancy,
* Severe extraarticular deformity,
* Posttraumatic and septic arthritis sequel

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Estimated)
Dates: Start 2020-04-25 (Estimated); Primary Completion 2023-04-25 (Estimated); Study Completion 2023-07-25 (Estimated)

PRIMARY OUTCOMES:
anterior patellar offset ratio | From the date of randimization until the final follow up of last patient, assessed up to 15 months
  The distance between the anterior cortex of the femur and the maximum peak at the anterior of the prosthesis is considered as an "anterior femoral offset".Sagittal patellar offset defined by us as the ratio of the anterior femoral offset to the remaining distance between the maximum anterior point of the patella and the posterior vertex in the direct lateral knee joint radiography.

CONTACTS AND LOCATIONS:
Overall Officials: Orkhan Aliyev, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Scott CEH, Clement ND, Yapp LZ, MacDonald DJ, Patton JT, Burnett R. Association Between Femoral Component Sagittal Positioning and Anterior Knee Pain in Total Knee Arthroplasty: A 10-Year Case-Control Follow-up Study of a Cruciate-Retaining Single-Radius Design. J Bone Joint Surg Am. 2019 Sep 4;101(17):1575-1585. doi: 10.2106/JBJS.18.01096. PMID 31483401
- [Background] Liu S, Long H, Zhang Y, Ma B, Li Z. Meta-Analysis of Outcomes of a Single-Radius Versus Multi-Radius Femoral Design in Total Knee Arthroplasty. J Arthroplasty. 2016 Mar;31(3):646-54. doi: 10.1016/j.arth.2015.10.017. Epub 2015 Oct 26. PMID 26614746